CLINICAL TRIAL: NCT04655105
Title: Evaluation of Post Operative Pain Following Reciprocating and Rotary Heat-treated NiTi Instrumentation of Root Canals: a Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tamil Nadu Dr.M.G.R.Medical University (Other)
Responsible Party: Principal Investigator, Valliappan CT, post graduate student, Tamil Nadu Dr.M.G.R.Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TamilNadu
Record Dates: First submitted 2020-12-03; First posted 2020-12-07 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Root Canal Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Truanatomy rotary file (Experimental): use of tru anatomy rotary files root canal instrumentation followed by post operative pain evaluation
  Interventions: Device: root canal rotary files
- hyflex EDM rotary file (Experimental): use of hyflex EDM rotary files root canal instrumentation followed by post operative pain evaluation
  Interventions: Device: root canal rotary files
- edge endo reciprocating rotary file (Experimental): use of edge endo reciprocating rotary files root canal instrumentation followed by post operative pain evaluation
  Interventions: Device: root canal rotary files
- protaper gold rotary file (Active Comparator): use of protaper gold rotary files root canal instrumentation followed by post operative pain evaluation
  Interventions: Device: root canal rotary files

INTERVENTIONS:
Device: root canal rotary files — post operative pain evaluation using different rotary file system

SUMMARY:
The present clinical evaluation was planned for comparing the post-operative pain incidence in maxillary premolar teeth with acute irreversible pulpitis treated by recently introduced heat treated TruNatomy TM and other widely studied heat-treated files Hyflex EDM, Protaper Gold and one heat-treated reciprocating EdgeFile in single-visit root canal treatment.

DETAILED DESCRIPTION:
Essential component of successful root canal treatment is removal of pulp tissue remnants, microorganisms, and microbial toxins from root canal system. Machine assisted root canal preparation allows for faster and easier instrumentation. Flexible nickel-titanium (NiTi) root canal files have become indispensible with technological advancements in metallurgy and incorporation of several design features manufacturers have attempted to improve the efficiency of these instruments. 1 Thermomechanically treated NiTi has a modified phase composition compared to conventional NiTi files. These files contain varying amounts of R-phase and martensite in their alloy composition in clinical conditions. Increased proportion of martensite phase allows for more flexible files with enhanced cyclic fatigue resistance. Simultaneously endodontic motor have undergone significant enhancements regarding torque control and kinematics that are adjustable in several directions. 1 Yared (2008) introduced the concept of single file reciprocation which was based on balanced-force technique. Reciprocation motion have been shown to increase the cyclic fatigue resistance of NiTi instruments, also these motions have been associated with increased debris extrusion and post treatment discomfort. Recently TruNatomy TM files has been introduced with manufacturers claims of 0.8mm slim wire NiTi design with superior flexibility, off-centered cross-section, special heat-treated NiTi wire and regressive taper allowing for preservation of dentin and tooth integrity.

Post operative pain following root canal treatment is influenced by number of factors; root canal file system and rotary kinetics on incidence and intensity of post-operative pain has been conflicting with certain evidence favoring full rotary motion whilst others recommend reciprocating motion. Sun et al. (2018) in their systematic review concluded that different type of full rotary root canal NiTi file system did not have significant influence on post-root canal treatment pain and reciprocation motion was associated with increased post treatment discomfort. These scientific studies involved comparing both conventional NiTi and heat-treated files.

In this scenario the present clinical evaluation was planned for comparing the post-operative pain incidence in maxillary premolar teeth with acute irreversible pulpitis treated by recently introduced heat treated TruNatomy TM and other widely studied heat-treated files Hyflex EDM, Protaper Gold and one heat-treated reciprocating EdgeFile in single-visit root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included maxillary premolars with radiograph evidence of decay approximating the pulp with sound periodontal health.

Exclusion Criteria:

* Exclusion criteria were patients not willing for recall visits, teeth not amenable to post-endodontic restoration, teeth with periapical radiolucencies, presence of additional roots or canal variations from conventional maxillary premolar anatomy, two or more adjacent teeth requiring root canal treatment, absence of occlusal contacts, premolars not sufficiently anaesthetized with 2 mL of local anesthetic solution, teeth with difficult canal anatomy (curvatures > 30°, radiograph evidence of pulp chamber and canal calcification, open apices) immunocomprimised patients, patients systemic ailments hindering single-visit root canal treatment and pregnant patients.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-05-03 (Estimated); Study Completion 2021-06-03 (Estimated)

PRIMARY OUTCOMES:
post operative pain evaluation using different rotary instruments: VAS score | at 24 hrs
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain
post operative pain evaluation using different rotary instruments: VAS score | at 48hrs
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain
post operative pain evaluation using different rotary instruments: VAS score | at 7 days
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain

SECONDARY OUTCOMES:
assessment of pain scale using different rotary instruments | through study completion, an average of 1 week
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain
comparing the pain scale experienced between male and female in VAS score | through study completion, an average of 1 week
  pain scale is evaluated using VISUAL ANALOG SCALE (VAS) score (1-10) 1 is minimum amount of pain experienced and 10 is maximum amount of pain experienced [1-3] mild pain , [4-7] moderate pain , [8-10] severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- CSI college of dental sciences and research, Madurai, Tamil Nadu, India